CLINICAL TRIAL: NCT05271448
Title: The Effect of Continuing or Discontinuing ACE-I/ARBs Therapy on the Incidence of Contrast-induced Nephropathy in Patients With Chronic Kidney Disease Undergoing Coronary Angiography; a Randomized Controlled Trial
Brief Title: Continuing or Discontinuing ACE/ARBs in Patients With Chronic Kidney Disease Undergoing Coronary Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: An-Najah National University (Other)
Responsible Party: Principal Investigator, Yunis Daralammouri, Assistant Professor, An-Najah National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ACEI/ARBs/CKD/CATH
Record Dates: First submitted 2022-01-15; First posted 2022-03-09 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Contrast-induced Nephropathy; Chronic Kidney Diseases; Ischemic Heart Disease
Keywords: Cardiac catherization; coronary angiography; Coronary angioplasty; chronic kidney disease; contrast induced nephropathy; ACEI; ARBs
MeSH Terms: conditions — Renal Insufficiency, Chronic; Myocardial Ischemia | interventions — Enalapril; Ramipril; Valsartan; candesartan; Losartan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients enrolled to the study were randomized into continuing or discontinuing (ACEI/ARBs) group. Care providers and investigators collected their data before and after the coronary angiography. The independent variable - continuing or discontinuing (ACEI/ARBs) - was coded into A or B groups, then data was sent to the outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continue ACEI or ARBs (Experimental): Randomized to continue on prescribed ACE1 or ARBs
  Interventions: Other: Continue ACEI or ARBs ( Enalapril , Ramipril , Valsartan , Candesartan, Losartan )
- Hold ACEI or ARBs (Active Comparator): Angiotensin converting enzyme inhibitor or angiotensin receptor blocker held >= 24 hours pre-cardiac catheterization and restarted post-catheterization after creatinine measurement (48-72 hours post)
  Interventions: Other: Hold ACEI or ARBs

INTERVENTIONS:
Other: Continue ACEI or ARBs ( Enalapril , Ramipril , Valsartan , Candesartan, Losartan ) — Randomized to continue on prescribed ACE1 or ARBs ( Enalapril 5, 10, 20 mg // Ramipril 2.5 , 5 mg // Valsartan 80 , 160 mg // Candesartan 8, 16 mg // Losartan 50 mg )
  Other Names: Continue ACEI or ARBs
  Arms: Continue ACEI or ARBs
Other: Hold ACEI or ARBs — Angiotensin converting enzyme inhibitor or angiotensin receptor blocker held at least 24 hours pre-cardiac catheterization and restarted 48-72 hours post-catheterization (after creatinine measurement)
  Other Name: Includes all ACEI inhibitors or ARBs
  Arms: Hold ACEI or ARBs

SUMMARY:
Contrast induced nephropathy (CIN) is a well-known possible complication of percutaneous coronary intervention (PCI) with an incidence varies from 3.3% to 14.5% in patients undergoing PCI.

Many previous randomized and non-randomized studies have shown very conflicting results regarding the use of ACE-Is prior to coronary angiography, and whether it decreases or increases the risk of CIN. The importance of this study is to help find an acceptable and reliable answer for the use of ACE-I/ARBs prior to cardiac catheterization.

This research aims to study the effect of withholding ACE-Is or ARBs on the incidence of contrast induced nephropathy in patients undergoing coronary angiography who have chronic kidney disease (GFR<60 ml/min/1.73 m2) and to help build evidence-based data and guidelines on the safety of continuing or withholding ACE-I/ARBs pre contrast administration.

DETAILED DESCRIPTION:
The study design is a Randomized Control Trial; it will be done on two groups of patients. The two groups are group A (continue ACE-I/ARBs) and group B (withhold ACE-I/ARBs).

The study will be conducted at the cardiology units at An-Najah National University's hospital (NNUH) in Nablus, Palestine.

Study population includes chronic kidney disease patients taking ACE-I or ARBs therapy and are undergoing elective coronary angiography.

Patients who will meet the inclusion criteria and have none of the exclusion criteria will be enrolled in the trial when the appointment of their procedure is set.

They will be randomly divided into two groups; group A (continue ACE-I or ARBs therapy) and group B (withhold ACE-I or ARBs therapy)using block randomization, each block consists of four participants.

Patients in the continuation group will take their regular ACE-I/ARBs on the day of the angiogram. Patients in the discontinuation group will be withheld from their ACEI or ARBs 24 h before cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

1. At least one month of continuous therapy with an ACEI or an ARBs and
2. Undergoing elective coronary angiography and
3. Have CKD stage3-4 (15≤GFR<60 ml/min/1.73 m2).

Exclusion Criteria:

1. Acute STEMI within 2 weeks
2. NYHA class IV heart failure by history
3. Administration of contrast load within the previous 6 days
4. acute renal failure (ARF) preceding coronary angiography
5. potassium level more than 5.0 meq/l
6. GFR <15 ml/min/1.73 m2
7. previous percutaneous cardiac catheterization within one month
8. Acute pulmonary edema
9. hemodynamically instability
10. uncontrolled hypertension
11. combination ACEI and ARB therapy
12. Cardiogenic shock
13. Sepsis
14. pregnancy
15. Age below 18 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Contrast induced nephropathy | 48 - 72 hours post-cardiac catheterization
  Contrast induced nephropathy (creatinine rise of ≥0.5 mg/dL or a relative increase ≥25%compared to the pre-randomization creatinine level) at 48-72hrs

SECONDARY OUTCOMES:
Serum creatinine level | 48 - 72 hours post-cardiac catheterization
  Change in serum creatinine at 48-72hrs
Number of Participants with Hyperkalemia | 48 - 72 hours post-cardiac catheterization
  Serum potassium increased to > 5.5 mg/dL at 48-72hrs
Creatinine clearance | 48 - 72 hours post-cardiac catheterization
  Change in Creatinine clearance at 48-72hrs
Death, Myocardial Infarction, Stroke, Congestive Heart Failure, dialysis, major bleeding, minor bleeding, hypertension, re-hospitalization at 48-72hrs | 48 - 72 hours post-cardiac catheterization
  Death, Myocardial Infarction, Stroke, Congestive Heart Failure, dialysis, major bleeding, minor bleeding, hypertension, re-hospitalization at 48-72hrs

CONTACTS AND LOCATIONS:
Overall Officials: Yunis A Daralammouri, asst. prof., Principal Investigator — An-Najah National University
Locations (1):
- An-Najah National University Hospital, Nablus, West Bank, Palestinian Territories